CLINICAL TRIAL: NCT03794102
Title: The Effects of Water Versus Saline on Absorption Rates and Visualization During Ureteroscopy
Brief Title: Water Versus Saline as Irrigation Fluid for Ureteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kenneth Ogan, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00005780
Record Dates: First submitted 2018-12-21; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Ureteral Stricture; Hydronephrosis; Urothelial Carcinoma; Urolithiasis
MeSH Terms: conditions — Hydronephrosis; Carcinoma, Transitional Cell; Urolithiasis | interventions — Water; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ureteroscopy with water irrigation (Active Comparator): Participants meeting medical requirements to undergo ureteroscopy will undergo a routine cystoscopy and ureteroscopy following standard techniques. Water will be used as the irrigation fluid during the ureteroscopy.
  Interventions: Other: Water
- Ureteroscopy with saline irrigation (Active Comparator): Participants meeting medical requirements to undergo ureteroscopy will undergo a routine cystoscopy and ureteroscopy following standard techniques. Saline will be used as the irrigation fluid during the ureteroscopy.
  Interventions: Other: Saline

INTERVENTIONS:
Other: Water — Sterile water irrigation from standard sterile water bags will be used during ureteroscopy. Pulsed irrigation of the irrigant fluid with hand-held syringes will be used in all cases according to standard practice in order to visualize the upper urinary tract during the ureteroscopy procedure.
  Arms: Ureteroscopy with water irrigation
Other: Saline — 0.9% saline irrigation from standard saline bags will be used during ureteroscopy. Pulsed irrigation of the irrigant fluid with hand-held syringes will be used in all cases according to standard practice in order to visualize the upper urinary tract during the ureteroscopy procedure.
  Arms: Ureteroscopy with saline irrigation

SUMMARY:
The purpose of this study is to determine the rate of absorption of fluids (water or saline) during ureteroscopy and to assess the effects on electrolyte levels. The investigators also want to measure how much better the urologist can see the ureter based on the type of irrigation fluid that is used.

DETAILED DESCRIPTION:
The use of fluid irrigation is important during urologic procedures. There is little research done on the use of water versus saline for irrigation during ureteroscopy.

This study will evaluate whether the use of water or saline during ureteroscopy has any clinical implications. The investigators will compare the amount of fluid absorbed and differences in electrolytes between the two participant groups.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Participants meeting medical requirements to undergo ureteroscopy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Amount of irrigation fluid used during ureteroscopy | Measurement will be performed day of ureteroscopy
  At conclusion of the ureteroscopy, the bag with the remaining fluid will be weighed to determine amount of fluid used. The study will last from the start to the completion of the ureteroscopy, i.e. the duration of the ureteroscopic evaluation.
Change in serum sodium levels | Measurement will be performed day of ureteroscopy
  Blood samples will be drawn preoperatively and at conclusion of case (prior to awakening the participant) to assess the serum sodium levels (mEq/L). The study will last from the start to the completion of the ureteroscopy, i.e. the duration of the ureteroscopic evaluation.
Surgeon's rating of ureteroscopic visualization | Measurement will be performed day of ureteroscopy
  The surgeon will be asked to rate the degree of ureteroscopic visualization on a scale of 1-5, where 1=Poor visualization and 5= Excellent visualization. The study will last from the start to the completion of the ureteroscopy, i.e. the duration of the ureteroscopic evaluation.
Measurement of fluid clarity | Measurement will be performed day of ureteroscopy
  Fluid clarity was assessed by taking turbidity (cloudiness) measurements of renal fluid (in nephelometric turbidity units (NTU)) with a turbidimeter. The average of three measurements of turbidity was used at the fluid clarity measurement of each case, to supplement the ureteroscopic visualization measurement by surgeon rating. The study will last from the start to the completion of the ureteroscopy, i.e. the duration of the ureteroscopic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ogan, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Emory University, Atlanta, Georgia